CLINICAL TRIAL: NCT04789915
Title: AMEND - Add-on MEmaNtine to Dopamine Modulation to Improve Negative Symptoms at First Psychosis
Brief Title: Add-on MEmaNtine to Dopamine Modulation to Improve Negative Symptoms at First Psychosis
Acronym: AMEND
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bjorn H. Ebdrup (Other)
Collaborators: Lundbeck Foundation (Other); Danish Research Centre for Magnetic Resonance (Other)
Responsible Party: Sponsor-Investigator, Bjorn H. Ebdrup, Professor, MD PhD, leader of CNSR, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-001061-20
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Psychosis; Negative Symptoms With Primary Psychotic Disorder
Keywords: Memantine; Aripiprazole; 7 tesla MR
MeSH Terms: conditions — Psychotic Disorders | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Memantine + aripiprazole (Active Comparator): Tablet memantine or placebo will be initiated at 10mg/day for 1 week, hereafter the dose will be increased to 20mg/day until end of trial. The tablets will be identical and be provided in 10mg tablets or 20 mg tablets. (12 weeks of treatment).
  Tablet aripiprazole will be administered in doses starting at 5-10 mg/day. Doses will be increased slowly according to effect and side effects up to 30 mg/day.
  Interventions: Drug: Memantine
- Placebo + aripiprazole (Placebo Comparator): Coated placebo tablets will be provided to match memantine. Placebo equivalent of 10mg/day for 1 week, hereafter the dose will be increased to 20mg/day until end of trial. (12 weeks of treatment).
  Tablet aripiprazole will be administered in doses starting at 5-10 mg/day. Doses will be increased slowly according to effect and side effects up to 30 mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Add on treatment with memantine to aripiprazole.
  Arms: Memantine + aripiprazole
Drug: Placebo — Placebo add on to aripiprazole
  Arms: Placebo + aripiprazole

SUMMARY:
Antipsychotics affects the brain's dopamine system, and the drugs reduce delusions, hallucinations, and disorganized thinking, which are cardinal symptoms of psychotic disorders. However, negative symptoms e.g. anhedonia, avolition, and social withdrawal, as well as cognitive deficits, are not sufficiently treated.

Memantine is used to treat Alzheimer's disease and affects the brain's glutamate system. AMEND is a 12-week, double-blind, placebo-controlled, randomized clinical trial (RCT) testing effects of add-on memantine to initial antipsychotic treatment in never-treated patients with first-episode psychosis.

The main aim is to reduce negative symptoms. Secondary outcomes are cognition, psychotic symptoms, side effects. Glutamate levels in the brain will be measured before and after 12 weeks using an ultra-high field strength (7 Tesla) magnetic resonance scanner.

AMEND will apply rational drug repurposing to optimize treatment of patients experiencing their first psychotic episode.

DETAILED DESCRIPTION:
BACKGROUND Scientific basis/Rationale Antipsychotic medication is efficacious in treating positive psychotic symptoms such as delusions, hallucinations, and disorganized thinking, which are cardinal symptoms of schizophrenia spectrum disorders. However, antipsychotic treatment does not ameliorate the accompanying negative symptoms (e.g. anhedonia, avolition, and social withdrawal), and cognitive deficits, which are highly disabling and predictive of patients' long-term prognosis. Importantly, shortening the interval between onset of psychosis and initiation of an efficient intervention lead to better long-term outcome.

The pathophysiology of psychosis is complex and involves multiple neurotransmitters, e.g. serotoninergic-, GABAergic, and glutamatergic systems, but modulation (particularly antagonism) of striatal dopamine D2 receptors (D2R) remain the key common denominator of all licensed antipsychotics. Nevertheless, around one third of patients with psychosis display inadequate response to antidopaminergic treatment, and persistent negative symptoms is a critical predictor for future treatment resistance.

Glutamate hypothesis of psychosis Mounting evidence from post-mortem-, brain imaging-, genetic-, and pharmacologic challenge studies indicate glutamatergic dysregulation, specifically of the N-methyl-D-aspartate receptor (NMDAR), as part of the pathophysiology of psychosis and schizophrenia. Through excitotoxicity, glutamate dysregulation may underlie structural degeneration, e.g. in hippocampus, which is a key finding in schizophrenia spectrum patients. Nevertheless, cross-sectional 3T MRS glutamate levels between first-episode patients and HC have shown equivocal results, e.g. likely reflecting differences in glutamate levels across brain regions and in variable previous antipsychotic exposure of included patients. Using 3T MRS, investigator recently reported increased thalamic glutamate levels in antipsychotic-naïve patients with first-episode psychosis compared to HC. Importantly, high thalamic levels predicted poor treatment response. Other studies have also associated glutamate levels with outcome. Investigator have shown that aberrations in the thalamic glutamate levels are heritable, related to psychosis, and extend to individuals at ultra-high risk for psychosis (UHR). Investigator have found that thalamic and ACC levels of glutamate are associated with symptomology and cognition, specifically spatial working memory, set-shifting, and attention both in UHR and first episode psychosis. Cutting-edge 7T MRS can non-invasively determine brain metabolite levels of e.g. γ-aminobutyric acid (GABA), N-acetylaspartate, N-acetylaspartyl, and importantly, 7T allows to discriminate glutamate concentrations from glutathione and glutamine. Moreover, multiple voxels/brain regions can be investigated with 7T. In the context of glutamate and psychosis, the thalamus, anterior cingulate cortex (ACC), hippocampus, dorsolateral prefrontal cortex (DLPFC), and basal ganglia are of particular interest.

Regarding brain structure, application of structural 7T sequences allows for increased sensitivity to quantify neurodegeneration e.g. hippocampal subfield segmentation. Finally, high resolution quantification of tissue parameters such as iron deposition using quantitative susceptibility mapping allow characterization of subtle changes in the 'dopaminergic regions' of the basal ganglia, including striatum, pallidum, and substantia nigra.

Glutamate antagonist treatment Against this background, modulation of glutamatergic NMDAR has been investigated as a potential treatment target in patients with psychosis and schizophrenia. Memantine is a non-competitive NMDAR antagonist used for treatment of Alzheimer's disease. Two recent meta-analyses and one systematic review have concluded that adjunctive memantine to antipsychotics is safe and significantly improves negative symptoms in chronic medicated patients with schizophrenia. One of the meta-analyses also indicated a potential effect on global levels of cognition. Memantine has been theorized to ameliorate progression of negative symptoms by counteracting excitotoxicity correlated to high glutamate levels in early stages of psychosis, but this has not been investigated in initially antipsychotic-naïve patients. Finally, the intriguing fact that pharmacologically similar antagonists of NMDARs (e.g. memantine and ketamine) exert almost paradoxical effects in humans highlights the importance of understanding the pathophysiology of NMDAR modulation in psychosis.

Study medication Aripiprazole Aripiprazole is a partial dopamine D2 receptor agonist, approved for treatment of schizophrenia and now recommended as first choice of treatment in young patients with debut of symptoms due to a more favorable side-effect profile, than other antipsyychotics. The mechanism of action is mediated through a combination of partial agonism at dopamine D2 and serotonin 5-HT1A receptors and antagonism of serotonin 5-HT2A receptors. Common side effects include blurred vision, akathisia, tremor, headache, anxiety and metabolic changes (se section on side effects for full list). We have previously used aripiprazole in a previous cohort and have MRI and PET data for relevant comparison.

Memantine Tablet memantine (10-20 mg/day) is an generic drug approved for treatment of Alzheimer's Disease(AD) showing benefits on the main domains of AD i.e. cognition, function, behavior, and clinical global change. Memantine acts through uncompetitive, open-channel NMDAR antagonism, and has minimal activity for GABAergic, dopaminergic, adrenergic, histaminergic, and glycinergic receptors. There are no known interactions between memantine and antipsychotics. Side effects include fatigue, dizziness, constipation, anxiety, headache, diarrhoea, and nausea. In previous memantine add-on RCTs in schizophrenia patients, the reported side effects did not differ from placebo. Memantine has no abuse potential.

Placebo Placebo tablets will be coated to match memantine 10 or 20 mg.

Study population Antipsychotic-free, first-episode schizophrenia spectrum patients with first-episode psychosis.

Patients will be recruited from psychiatric hospitals and outpatients psychiatric centers in the capital region (Copenhagen area), where doctors or nursing staff will inform relevant patients about the project and contact the doctor or nurse from the AMEND team, if the patients accept and might fulfil the inclusion criteria. A diagnostic interview, Present State Examination(PSE), will be performed before inclusion to assess if the patients fulfil the inclusion criteria. In addition, to fulfilling the diagnostic criteria, it should be medically assessed that the patient would benefit from antipsychotic treatment. Furthermore, somatic and neurological examination, as well as screening of pregnancy and substance abuse, will be performed before inclusion.

Aim of study/ outstanding research questions to be answered in our study? Summary of concept By rational combination of two licensed, off-patent drugs, aripiprazole and memantine, AMEND aims to optimize treatment of psychosis alongside with unravelling the signature of memantine response. If successful, AMEND will provide pivotal neurobiological evidence for future stratification of patients with first-episode psychosis before initial antipsychotic treatment.

Hypotheses

Investigator hypothesize that add-on of memantine to aripiprazole:

* Will be superior to reduce negative symptoms and that this effect will correlate with reduced glutamate levels in thalamus after 12 weeks.
* Will exert the most pronounced effect in patients, who display higher baseline thalamic glutamate levels than HC, and this subgroup of patients will also experience better total symptom control.
* Will improve domains of cognition, and specifically that effects on working memory, set-shifting, and attention will be predicted by initial glutamate levels in thalamus and anterior cingulate cortex (ACC).

Primary and secondary endpoints Primary Endpoints Primary endpoint will be reduction in negative symptoms as measured with Positive and Negative Syndrome Scale (PANSS) negative symptoms after 12 weeks of treatment [PANSS negative baseline - PANSS negative at week 12]. Assessments will be supplemented by Brief Negative Symptom Scale (BNSS) scores.

Secondary endpoints Secondary endpoints include changes in cognition (in particular working memory, set-shifting, and attention), PANSS positive and total other clinical measures, level of functioning, side effects, and glutamate levels in five a priori selected regions: thalamus, anterior cingulate cortex (ACC), hippocampus, dorsolateral prefrontal cortex (DLPFC), and basal ganglia.

Exploratory endpoints include associations between clinical data, quality of life, brain metabolites in other regions, e.g. ACC, and structural measures (e.g. hippocampus subfields), and basal ganglia quantification. Interactions between baseline brain metabolite levels and brain structure in patients and HC will also be investigated.

Material and methods Study design This investigator-initiated, double blinded randomized controlled trial, will establish a cohort of 46 antipsychotic- free first episode psychosis patients aged 18-45. Patients will be recruited from psychiatric out- and inpatient clinics in the Capital Region of Copenhagen.

Patients will be allocated to 12 weeks treatment with [aripiprazole plus memantine] OR [aripiprazole plus placebo]. Randomisation will be stratified by PANSS negative sub score categorizing patients in a "Low PANSS baseline<20" and "High PANSS baseline>=20".

The randomisation will use permuted blocs in sizes of 4,6 and 8, to ensure an even distribution among the two groups since the number of patients in the two groups will not be restricted.

The pharmacy (Region Hovedstadens apotek) will manage the randomisation. Twenty healthy controls matched on age, gender and parental socio-economic status will be recruited by advertisement and undergo baseline- and 12-week examinations.

Trial design Double blinded randomized controlled trial.

Study phase Phase I, known medicine (memantine) tested for new indication (psychosis).

Timeline Estimated study duration To increase power of secondary analyses, enrolment will continue until 18 participants in each arm have completed examinations. Moreover, AMEND will be extended to 12 weeks based on the median trial duration in the meta-analysis of add-on memantine (12 weeks (mean 11.5 weeks)).

Based on our center's 20 years of experience with recruitment and treatment of antipsychotic-free patents, we expect an inclusion rate of 2 patients per month and an attrition rate of 25%. Thus, recruitment of 46 patients will take 2 years.

Amendment to the protocol, march 2023:

We have converted the antipsychotic used in the study from amisulpride to aripiprazole. Originally amisulpride was chosen - among several recommended antipsychotic options - based on a pharmacological argument (selectivity for the dopamine D2/3 receptor). However, since the protocol was written and approved, the treatment guideline has been updated. After the update, the first line treatment for psychotic patients, who have never been treated before is now aripiprazole due to fewer side effects.

Understandably, the update has given rise to reluctancy from clinicians to refer patients to a study using a treatment which is no longer first-line. As a consequence, we have observed a decline in referrals and within the referred group a remarkably high proportion of patients with schizophrenia simplex, which is a rather rare condition not representative of the general patient with first-episode psychosis.

To further increase requitement and feasibility we modify the exclusion criterion: "Never medicated with antipsychotic medicine", to now accept patients who previously have been minimally exposed to antipsychotic medication. We apply the criteria used in the large European OPTiMiSE trial.

Our power calculation is based on detecting a small clinical difference between the two groups (2 points in PANSS negative symptoms). Therefore, we are sensitive with regard to analyzing a representative sample of the study population. In addition, we are applying for permission to extend the cohort, so we can continue to include patients until 36 patients has completed the study program with aripiprazole + (memantine/placebo) as treatment.

In the AMEND study, the basic question is to test the effect of add-on memantine to an antipsychotic drug and not to specifically test the effect of add-on memantine to amisulpride per se. We consider it of utmost importance to retain high clinical value of AMEND. Therefore, we consider is ethically sound to propose these two modifications (change to aripiprazole and minimally mediation prior to inclusion) to the AMEND protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Antipsychotic-free(as defined under Exclusion Criteria below), first episode psychosis
  * Fulfilling the diagnostic criteria of schizophrenia, persistent delusional disorder, acute and transient psychotic disorders, schizoaffective disorder, other non-organic psychotic disorders and unspecified non-organic disorders (ICD-10: F20.x; F22.x; F23.x; F24.x; F25.x; F28; F29); verified by PSE interview.
  * Age: 18-45 years
  * Legally competent (In Danish: 'myndige og habile i retslig forstand')

Healthy controls:

* No first-degree relative with known major psychiatric disorder (ICD-10: F1x; F2x; F3x)
* Age 18-45 years
* Legally competent (In Danish: 'myndige og habile i retslig forstand')

Exclusion Criteria:

* Patients

  * Prior use of antipsychotic medication longer than an episode of two weeks in the previous year and/or 6 weeks lifetime, and/or antipsychotic treatment within 30 days prior to inclusion.
  * Treatment with antidepressant medication the last 7 days
  * Current substance dependence ICD-10 (F1x.2) or substance abuse in any period up to 3 months prior to referral (exception: tobacco/nicotine, F17.2)
  * Head injury with more than 5 minutes of unconsciousness, lifetime
  * Any coercive measure
  * Metal implanted by operation
  * Head or neck tattoos
  * Pacemaker
  * Pregnancy (assessed by urine HCG)
  * Female patients: Unwillingness to use safe contraception (Intra Uterine Device/System or hormonal contraceptives) during the study period.
  * Severe physical illness
  * Allergies to any of the ingredients in the aripiprazole tablets or memantine tablets

Healthy controls:

* Lifetime substance abuse/dependence ICD-10 (F1x.1/F1x.2) (exception: tobacco/nicotine, F17.1/F17.2)
* Lifetime treatment with antidepressants
* Head injury with more than 5 minutes of unconsciousness
* Metal implanted by operation
* Head or neck tattoos
* Pacemaker
* Pregnancy (assessed by urine HCG)
* Severe physical illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative Symptom change, PANSS negative subscore | 12 weeks
  Change in negative symptoms measured on the Positive and negative syndrome scale (PANSS), negative symptom subscore total. Scale from 7 to 49, lower values indicating better outcome.
Negative Symptom change, Brief Negative Symptom Scale (BNSS) | 12 weeks
  Change in negative symptoms measured on the Brief Negative Symptom Scale (BNSS).
  Scale from 0 to 90, lower values indicating better outcome.

SECONDARY OUTCOMES:
PANSS total | 12 weeks
  Overall clinical effect measured on Positive and negative syndrome scale (PANSS) total.
  Scale from 30 to 210, lower values indicating better outcome.
PANSS positive | 12 weeks
  Change in positive symptoms measured on the Positive and negative syndrome scale (PANSS), positive symptom subscore total.
  Scale from 7 to 49, lower values indicating better outcome.
Cognition, CANTAB | 12 weeks
  Change in cognitive measurements:
  Cambridge Neuropsychological Test Automated Battery (CANTAB)
Cognition, BACS | 12 weeks
  Change in cognitive measurements:
  Brief Assessment of Cognition in Schizophrenia (BACS): memory, working memory, processing speed, executive functions and verbal fluency
MR spectroscopy 1 | 12 weeks
  7 tesla MR scan with spectroscopy seqcuenses. Glutamate levels in thalamus
MR spectroscopy 2 | 12 weeks
  7 tesla MR scan with spectroscopy seqcuenses. Glutamate levels in anterior cingulate cortex (ACC)
MR spectroscopy 3 | 12 weeks
  7 tesla MR scan with spectroscopy seqcuenses. Glutamate levels in hippocampus
MR spectroscopy 4 | 12 weeks
  7 tesla MR scan with spectroscopy seqcuenses. Glutamate levels in dorsolateral prefrontal cortex (DLPFC)
MR spectroscop5 | 12 weeks
  7 tesla MR scan with spectroscopy seqcuenses. Glutamate levels in the basal ganglia

OTHER OUTCOMES:
Quality of life, self rated by patients | 12 weeks
  Measured on quality of life scale (QLS), by patients. Scale with 21 items, from 0 to 4, total scores from 0 to 84. Higher scores indicating a better quality of life.
MR exploratory outcomes, spectroscopy | 12 weeks
  Spectroscopy data (glutamate and GABA concentrations) from other regions
MR exploratory outcomes, structural data 1 | 12 weeks
  MR structural measurements, volumetric data of thalamus
MR exploratory outcomes, structural data 2 | 12 weeks
  MR structural measurements, volumetric data of anterior cingulate cortex (ACC)
MR exploratory outcomes, structural data 3 | 12 weeks
  MR structural measurements, volumetric data of hippocampus
MR exploratory outcomes, structural data 4 | 12 weeks
  MR structural measurements, volumetric data of dorsolateral prefrontal cortex (DLPFC)
MR exploratory outcomes, structural data 5 | 12 weeks
  MR structural measurements, volumetric data of the basal ganglia

CONTACTS AND LOCATIONS:
Overall Officials: Olga B Baltzersen, MD, Principal Investigator — CNSR, Metal Health Centre Glostrup
Locations (1):
- Centre for Neuropsychiatric Schizophrenia Research, CNSR & Centre for Clinical Intervention & Neuropsychiatric Schizophrenia Research, CINS, Glostrup Municipality, Capitol Region, Denmark

REFERENCES:
- [Derived] Sandstrom KO, Baltzersen OB, Marsman A, Lemvigh CK, Boer VO, Bojesen KB, Nielsen MO, Lundell H, Sulaiman DK, Sorensen ME, Fagerlund B, Lahti AC, Syeda WT, Pantelis C, Petersen ET, Glenthoj BY, Siebner HR, Ebdrup BH. Add-On MEmaNtine to Dopamine Antagonism to Improve Negative Symptoms at First Psychosis- the AMEND Trial Protocol. Front Psychiatry. 2022 May 20;13:889572. doi: 10.3389/fpsyt.2022.889572. eCollection 2022. PMID 35669271